CLINICAL TRIAL: NCT03973333
Title: A Phase 1/2 First-in-human Study of the Safety and Efficacy of IMC-C103C as Single Agent and in Combination With Atezolizumab in HLA-A*0201-positive Patients With Advanced MAGE-A4-positive Cancer
Brief Title: Safety and Efficacy of IMC-C103C as Monotherapy and in Combination With Atezolizumab
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study withdrawn by Sponsor
Sponsor: Immunocore Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IMC-C103C-101
Record Dates: First submitted 2019-05-23; First posted 2019-06-04 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Select Advanced Solid Tumors
Keywords: ImmTAC, IMC-C103C, MAGE-A4, immunotherapy
MeSH Terms: interventions — atezolizumab

STUDY DESIGN:
Intervention Model Description: Sequential from arm monotherapy IV dose escalation is opened first; then monotherapy SC dose escalation, monotherapy expansion and combination dose escalation may run
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- IMC-C103C - Monotherapy IV dose escalation (Experimental): n= approximately 50 patients to establish the MTD/expansion dose
  Interventions: Drug: IMC-C103C
- IMC-C103C and atezolizumab dose escalation (Experimental): n=approximately 12 patients to establish the MTD/expansion dose
  Interventions: Drug: IMC-C103C; Drug: Atezolizumab
- IMC-C103C - expansion (Experimental): Patients will be enrolled n=9-24 per expansion cohort (up to 4 total): metastatic/unresectable tumors of interest patients treated at the expansion dose of IMC-C103C to assess preliminary anti-tumor efficacy
  Interventions: Drug: IMC-C103C
- IMC-C103C monotherapy SC dose escalation (Experimental): Patients will be enrolled n=9-12 to establish the MTD/expansion dose
  Interventions: Drug: IMC-C103C

INTERVENTIONS:
Drug: IMC-C103C — Weekly IV infusions
  Arms: IMC-C103C - Monotherapy IV dose escalation; IMC-C103C - expansion; IMC-C103C and atezolizumab dose escalation
Drug: Atezolizumab — IV infusions every 3 weeks
  Other Names: TECENTRIQ
  Arms: IMC-C103C and atezolizumab dose escalation
Drug: IMC-C103C — Weekly subcutaneous Injection
  Arms: IMC-C103C monotherapy SC dose escalation

SUMMARY:
IMC-C103C is an immune mobilizing monoclonal T cell receptor against cancer (ImmTAC ®) designed for the treatment of cancers positive for the tumor-associated antigen MAGE-A4. This is a first-in-human trial designed to evaluate the safety and efficacy of IMC-C103C in adult patients who have the appropriate HLA-A2 tissue marker and whose cancer is positive for MAGE-A4.

DETAILED DESCRIPTION:
The IMC-C103C-101 Phase 1/2 study will be evaluated in patients with metastatic/unresectable tumors which include select Advanced Solid Tumors and will be conducted in two phases.

1. To identify the maximum tolerated dose (MTD) and/or expansion dose of IMC-C103C as a single agent administered intravenously (IV) and subcutaneously (SC) once weekly (Q1W) and administered Q1W in combination with once every 3 weeks (Q3W) atezolizumab.
2. To assess the preliminary anti-tumor activity of IMC-C103C in one or more selected indications, as a single agent administered Q1W.

ELIGIBILITY:
Inclusion Criteria:

1. HLA-A*02:01 positive
2. MAGE-A4 positive tumor
3. Eastern Cooperative Oncology Group (ECOG) performance status (PS) [ECOG PS] 0 or 1
4. Selected advanced solid tumors
5. Relapsed from, refractory to, or intolerant of standard therapy
6. Measurable disease per RECIST v1.1 (expansion)
7. If applicable, must agree to use highly effective contraception

Exclusion Criteria:

1. Symptomatic or untreated central nervous system metastasis
2. Inadequate washout from prior anticancer therapy
3. Significant ongoing toxicity from prior anticancer treatment
4. Impaired baseline organ function as evaluated by out-of-range laboratory values
5. Clinically significant cardiac disease
6. Active infection requiring systemic antibiotic therapy
7. Known history of human immunodeficiency virus (HIV)
8. Active hepatitis B virus (HBV) or hepatitis C virus (HCV)
9. Ongoing treatment with systemic steroids or other immunosuppressive therapies
10. Significant secondary malignancy
11. Pregnancy or lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-05-17 (Estimated); Primary Completion 2023-09-25 (Estimated); Study Completion 2023-09-25 (Estimated)

PRIMARY OUTCOMES:
Phase 1: Incidence of dose-limiting toxicities (DLT) | From first dose to DLT period (28 days)
Phase 1: incidence and severity of adverse events (AE) | from first dose to 30 days after the last dose
Phase 1: changes in laboratory parameters | from first dose to 30 days after the last dose
  Abnormalities will be classified according to NCI CTCAE v5.0
Phase 1: changes in vital signs | from first dose to 30 days after the last dose
  Abnormalities will be classified according to NCI CTCAE v5.0
Phase 1: changes in electrocardiogram parameters | from first dose to 30 days after the last dose
  QT intervals corrected for heart rate using Fridericia's (cube root) correction (QTcF) interval absolute values and changes from baseline will be summarized
Phase 1: dose interruptions, reductions, and discontinuations | from first dose through last dose (anticipated for up to 12-24 months)
Phase 2: Best overall response (BOR) | from first dose to approximately 2 years

SECONDARY OUTCOMES:
Phase 2: incidence and severity of adverse events (AE) | from first dose to 30 days after the last dose
Phase 2: changes in laboratory parameters | from first dose to 30 days after the last dose
  Abnormalities will be classified according to NCI CTCAE v5.0
Phase 2: changes in vital signs | from first dose to 30 days after the last dose
  Abnormalities will be classified according to NCI CTCAE v5.0
Phase 2: changes in electrocardiogram parameters | from first dose to 30 days after the last dose
  QTcF interval absolute values and changes from baseline will be summarized
Phase 2: dose interruptions, reductions, and discontinuations | from first dose through last dose (anticipated for up to 12-24 months)
Phase 1: Best overall response | from first dose to approximately 2 years
Progression-free survival | from first dose to approximately 2 years
Duration of response | from first dose to approximately 2 years
Overall survival | from first dose to approximately 2 years
Pharmacokinetics Area under the plasma concentration-time curve (AUC) | from first dose to within approx, 2 weeks of last dose/4 weeks (IMC-C103C AUC will be assessed weekly for 4 weeks)
Pharmacokinetics The maximum observed plasma drug concentration after single dose administration (Cmax) | from first dose to within approx, 2 weeks of last dose/4 weeks (IMC-C103C AUC will be assessed weekly for 4 weeks)
Pharmacokinetics The time to reach maximum plasma concentration (Tmax) | from first dose to within approx, 2 weeks of last dose/4 weeks (IMC-C103C AUC will be assessed weekly for 4 weeks)
Pharmacokinetics The elimination half-life (t1/2) | from first dose to within approx, 2 weeks of last dose/4 weeks (IMC-C103C AUC will be assessed weekly for 4 weeks)
Immunogenicity the incidence of anti-drug antibody formation | from first dose to 14 days after the last dose
Changes in lymphocyte counts over time | from first dose to approx 4 weeks
Changes in serum cytokines over time | from first dose to approx.. 4wks
GCIG CA-125 response (ovarian carcinoma) | from first dose to approx.. 30 days after the last dose

CONTACTS AND LOCATIONS:
Locations (19):
- United States (10):
  - The Angeles Clinic and Research Institute, Los Angeles, California
  - University of California Davis Comprehenvise Cancer Center, Sacramento, California
  - University of Colorado Cancer Center, Aurora, Colorado
  - The University of Chicago Medicine & Biological Sciences, Chicago, Illinois
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Oklahoma University Medical Center, Oklahoma City, Oklahoma
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - UPMC Cancer Center, Pittsburgh, Pennsylvania
  - Sarah Cannon Research Institute at Tennessee Oncology, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
- Spain (4):
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Clinica Universidad Navarra, Madrid
  - Hospital Universitario La Paz - PPDS, Madrid
  - Clinica Universidad Navarra, Pamplona
- United Kingdom (5):
  - Beatson West of Scotland Cancer Centre, Glasgow, Scotland
  - The Clatterbridge Hospital Cancer Center, Bebington
  - Sarah Cannon Research Institute, London
  - The Christie NHS Foundation Trust, Manchester
  - Royal Marsden Hospital, Sutton